CLINICAL TRIAL: NCT06597968
Title: Performance Estimation of Triaging Artificial Intelligence Based Computer-Aided Detection Algorithm in Routine Chest Radiography
Brief Title: Evaluating the Real World Performance of an AI Based Lung Nodule Detection Tool
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Amit Gupta, MD, Associate Professor, Department of Radiology, School of Medicine Member, Cancer Imaging Program, Case Comprehensive Cancer Center, Cardiothoracic Division Chief department of Radiology, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20240362
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Nodule
Keywords: chest x-ray; CAD software

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Image going through AI tool: these are the images going through the AI tool
  Interventions: Device: AI Based CAD Software (qXR-Ln)
- image not going through AI tool: these are the images not going through the AI tool

INTERVENTIONS:
Device: AI Based CAD Software (qXR-Ln) — All x-ray images have already been obtained and will then be run through CAD software for secondary nodule detection
  Groups: Image going through AI tool

SUMMARY:
chest x-rays will be analyzed by AI software for a secondary read of lung nodules. Chest x-rays will either be sent to the AI tool to be read or to radiologists to read. If the image is sent to the AI tool, the AI software will generate a report on if it detects a lung nodule or not. The image will then be sent to a radiologist to determine if there is agreement or disagreement with the AI tool.

DETAILED DESCRIPTION:
The study is a prospective study for measuring the performance of an AI software in detecting lung nodules from chest X-rays. Data collected during the study will be analyzed for study purposes after end date of data collection.

There will be two study arms: the control arm and the interventional arm.

Control Arm:

There will be no interruption to the existing standard of care pathway.

Interventional Arm:

Use of AI will occur in parallel to the standard of care pathway.

Consistent with the control Arm, the radiologists or clinicians interpreting the chest x-ray images will proceed as usual based on the existing standard operating procedures of the study site. In addition, the AI software will function as a second reader; meaning images will be processed by the AI software which will generate a report.

In the event that the radiologist and the AI tool do not agree, cases will be reviewed by qualified study team members twice per week.

ELIGIBILITY:
Inclusion Criteria:

* Chest X-ray images of patients aged 18 - 89 years.
* Modality: CR/DR/DX.
* PA/view
* Lung nodules measuring 6 mm -30 mm (for chest X-ray images where presence of nodules is required).

Exclusion Criteria:

* Incomplete view of the chest.
* Lateral view
* Known lung cancer at the time of Chest x-ray images.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chest x-rays collected on patients aged 18-89
Sampling Method: Probability Sample
Enrollment: 45991 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
number of patients with actionable lung nodule as measured by CT scan | up to one year
total number of patients having chest x-ray | up to one year
number of patients with high risk lung nodule as measured by CT scan | up to one year
total number of patients referred for a CT scan | up to one year
number of lung nodule positive images | up to one year
number of lung nodule negative images | up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Amit Gupta, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No